CLINICAL TRIAL: NCT04996303
Title: Efficacy of Steroid Pulse Therapy in Acute Exacerbation of Idiopathic Pulmonary Fibrosis (AE-IPF) Admitted in ER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2021-0746
Record Dates: First submitted 2021-08-02; First posted 2021-08-09 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Idiopathic Pulmonary Fibrosis With Acute Exacerbation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine (Other): Routine steroid administration group
  Interventions: Drug: Routine steroid administration group
- Pulse (Other): Steroid pulse therapy group
  Interventions: Device: Steroid pulse therapy group

INTERVENTIONS:
Drug: Routine steroid administration group — Steroid administration with routine dose - Methylprednisolone 1 mg/kg 7 days → 0.5 mg/kg 7 days → 0.25 mg kg 7 days
  Arms: Routine
Device: Steroid pulse therapy group — Steroid administration with pulse dose - Methylprednisolone 10 mg/Kg (500 mg ~ 1g) pulse 3 days -> Methylprednisolone 1 mg/kg 7 days → 0.5 mg/kg 7 days → 0.25 mg/kg 7 days
  Arms: Pulse

SUMMARY:
Idiopathic pulmonary fibrosis is the most severe form of interstitial lung disease. It is known that the prognosis is poor due to extensive inflammation and fibrosis of the lung parenchyma. In case of acute exacerbation, the prognosis becomes worse. In early studies, the 3-month mortality rate reached 50-80%, and in a recent study, the 1-month survival rate was 66%, and the 3-month survival rate was 41%.

It is known that 20% of patients with IPF will experience acute exacerbations in their lifetime. The most commonly used treatment for such acute exacerbations is antibiotics and high-dose steroids, or steroid pulse therapy. However, its effectiveness is unclear, and the survival rate is still low. However, as there is no evident therapeutic agent other than steroids, it is included in the treatment guidelines, so conservative treatment is administered while steroids are administered to patients with acute exacerbation of idiopathic pulmonary fibrosis in most upper institutions.

There is no precise treatment other than steroids for patients with idiopathic pulmonary fibrosis-acute exacerbation, but the side effects of steroid administration cannot be overlooked. Therefore, a study is needed to confirm whether steroid pulse therapy is necessary or not.

1. Inclusion criteria

   * Among patients with clinically or histologically confirmed idiopathic pulmonary fibrosis, patients who visited the emergency room with dyspnea symptoms
   * Patients within 1 month of exacerbation of respiratory symptoms
   * Patients with increased GGO or worsening of IPF on chest CT within the last 2 weeks
   * Patients who understand the purpose of the clinical study and voluntarily agree to participate in this clinical study
   * When it is determined that steroid administration is necessary under the judgment of the medical staff during the treatment process
2. Exclusion criteria

   * Patients who complain of dyspnea symptoms due to causes other than the respiratory system, such as fluid overload, congestive heart failure, pulmonary embolism, etc.
   * Patients whose respiratory symptoms have worsened for more than 1 month
   * Persons who cannot read consent forms (eg. illiterate, foreigners, etc.)
3. Study design Using an open-label RCT randomization method, the administration will be divided into Group 1 (high-dose followed by low-dose steroid administration) and Group 2 (high-dose/low-dose steroid administration after steroid pulse therapy).

   * Test group: Group 1 (high dose followed by low dose steroid administration)
   * Control group: Group 2 (high-dose/low-dose steroid administration after steroid pulse therapy) ▶ Steroid administration Protocol Group 1: Methylprednisolone 1 mg/kg 7 days → 0.5 mg/kg 7 days → 0.25 mg kg 7 days Group 2: Methylprednisolone 10 mg/Kg (500 mg ~ 1g) pulse 3 days -> Methylprednisolone 1 mg/kg 7 days → 0.5 mg/kg 7 days → 0.25 mg/kg 7 days

Response evaluation

1. The level of inflammatory markers
2. Imaging improvement: chest x-ray or CT
3. Pulmonary function test: performed at the outpatient clinic before discharge or 12 weeks after the first visit for acute exacerbation

ELIGIBILITY:
Inclusion Criteria:

* Among patients with clinically or histologically confirmed idiopathic pulmonary fibrosis, patients who visited the emergency room with dyspnea symptoms
* Patients within 1 month of exacerbation of respiratory symptoms
* Patients with increased GGO or worsening of IPF on chest CT within the last 2 weeks
* Patients who understand the purpose of the clinical study and voluntarily agree to participate in this clinical study
* When it is determined that steroid administration is necessary under the judgment of the medical staff during the treatment process

Exclusion Criteria:

* Patients who complain of dyspnea symptoms due to causes other than the respiratory system, such as fluid overload, congestive heart failure, pulmonary embolism, etc.
* Patients whose respiratory symptoms have worsened for more than 1 month
* Persons who cannot read consent forms (eg. illiterate, foreigners, etc.)

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-07-18 (Actual)

PRIMARY OUTCOMES:
mortality rate | 3 months
  mortality rate depending on the steroid dose will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Moo Suk Park, Principal Investigator — Division of Pulmonology, Department of Internal Medicine, Severance Hospital, Yonsei University College of Medicine
Locations (1):
- Division of Pulmonology, Department of Internal Medicine, Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
The IPD could be shared with other researchers, including ILD specialists, especially laboratory data and underlying diseases.